CLINICAL TRIAL: NCT07327268
Title: Cyclic On-off Switching of Pulmonary Blood Flow in Moderate to Severe ARDS Patients With Mechanical Ventilation
Brief Title: Cyclic On-off Switching of Pulmonary Blood Flow in Moderate to Severe ARDS
Status: Not yet recruiting | Type: Observational
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Ling Liu, Principal Investigator, Southeast University, China
Other Study IDs: 3D-EIT perfusion
Record Dates: First submitted 2025-12-25; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: ARDS (Acute Respiratory Distress Syndrome); Electrical Impedance Tomography (EIT); Pulmonary Perfusion
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- phase 1: patients ventilated with a tidal volume of 4ml/kg pbw
- phase 2: patients ventilated with a tidal volume of 6ml/kg pbw
- phase 3: patients ventilated with a tidal volume of 8ml/kg pbw

SUMMARY:
Although the theoretical model of "cyclic on-off switching of pulmonary blood flow" provides a crucial perspective for understanding VILI, its clinical validation and real-time intervention face significant obstacles. The fundamental reason lies in the lack of pulmonary microcirculation monitoring technology capable of bedside, non-invasive, continuous operation with sufficient spatiotemporal resolution. Nowadays, a novel 3D-EIT can perform real-time and non-invasive assessment of the distribution of pulmonary blood flow. However, if 3D-EIT can help to identify "cyclic on-off switching of pulmonary blood flow" is still unclear.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients with mechanical ventilation
2. diagnosis of moderate to severe ARDS no more than 72 hours

Exclusion Criteria:

1. Chronic respiratory diseases that required long-term oxygen therapy, such as pulmonary fibrosis or chronical obstructive pulmonary disease
2. Contraindications to EIT (e.g., active implantable device, chest malformation, unstable spinal injuries or fractures, and open chest wounds)
3. Undrained pneumothorax or pneumomediastinum,
4. Hemodynamic instability
5. Pregnancy
6. Refusal by family or the attending physician to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients admitted to our ICU were screened for inclusion and exclusion criteria
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
The percent of "Cyclic On-Off Switching" | 15min
  "Cyclic On-Off Switching" was assessed by 3D-EIT

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda Hospital, School of Medicine, Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided